CLINICAL TRIAL: NCT01224587
Title: Characterisation of Gastrointestinal Transit of Four New Developed Gel Matrix Tablets With Different Erosion Rates by Means of MMM Measurement Under Fasting and Fed Conditions
Brief Title: Magnetic Marker Monitoring (MMM) Study With Gel Matrix Tablets Under Fasting and Fed Conditions
Acronym: MMM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1840M00017
Record Dates: First submitted 2010-10-12; First posted 2010-10-20 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Magnetic Marker Monitoring; Gastrointestinal-transport; Gastric Emptying Time; Small Intestinal Transit Time; Time for Colon Arrival; Food Effect
Keywords: Imaging technique; gastric transport through the gut

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): D1000078 placebo gel matrix tablet marked with approx. 5 mg Fe3O4(E172),AstraZeneca,Mölndal, Sweden , under fasting condition
  Interventions: Drug: D1000078
- 2 (Experimental): D1000082 placebo gel matrix tablet marked with approx. 5 mg Fe3O4(E172), AstraZeneca,Mölndal, Sweden, under fasting condition
  Interventions: Drug: D1000082
- 3 (Experimental): D1000083 placebo gel matrix tablet marked with approx. 5 mg Fe3O4(E172), AstraZeneca,Mölndal, Sweden ,under fasting condition
  Interventions: Drug: D1000083
- 4 (Experimental): D1000085 placebo gel matrix tablet marked with approx. 5 mg Fe3O4(E172), AstraZeneca,Mölndal, Sweden , under fasting condition
  Interventions: Drug: D1000085
- 5 (Experimental): D100083 marked with approx. 5 mg Fe3O4(E172), AstraZeneca,Mölndal, Sweden, under fed condition
  Interventions: Drug: D1000083
- 6 (Experimental): D1000085 placebo gel matrix tablet marked with approx. 5 mg Fe3O4(E172), AstraZeneca, Mölndal, Sweden , under fed condition
  Interventions: Drug: D1000085

INTERVENTIONS:
Drug: D1000078 — Oral, one single dose
  Arms: 1
Drug: D1000082 — Oral, one single dose
  Arms: 2
Drug: D1000083 — Oral, one single dose
  Arms: 3; 5
Drug: D1000085 — Oral, one single dose
  Arms: 4; 6

SUMMARY:
The purpose of this study is to monitor the gastrointestinal transport of eroding gel matrix placebo tablets in healthy male volunteers under fasting and fed conditions. The method which is used is an imaging technique.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic origin: Caucasian
* Body-mass index (BMI): ≥ 19 kg/m² and ≤ 27 kg/m²
* Good health
* Written informed consent, after having been informed about benefits and potential risks of the trial

Exclusion Criteria:

* Diseases which could influence the gastric emptying and gastrointestinal transport
* Diet which could influence the gastric emptying and gastrointestinal transport
* Surgery in the gastrointestinal tract which may interfere with the safety and transport of test product
* Ferromagnetic implants or any other magnetic disturbance, which can affect the Magnetic Marker Monitoring measurement
* Regular medical treatments which could affect the gastric emptying and gastrointestinal transport

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The time from an administration of each of the placebo gel matrix tablets of each arm until Gastric Emptying Time (GET)
The time from an administration of each of the placebo gel matrix tablets of each arm until Colon Arrival Time (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — Socra Tec R&D GmbH, Clinical Pharmacology Unit; Maria Anschütz, Study Chair — Socra Tec R&D GmbH
Locations (1):
- Research Site, Berlin, Germany